CLINICAL TRIAL: NCT00534742
Title: A Family-based Ischemic Stroke Study on Association and Interactions of Multi-pathway Genetic Polymorphisms
Brief Title: Fangshan / Family-based Ischemic Stroke Study In China
Acronym: FISSIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: National Natural Science Foundation of China (Other Government); Ministry of Education, China (Other Government); Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Principal Investigator, Yonghua Hu, Executive Dean, Peking University
Other Study IDs: NSFC-30671807; SRFDP-20060001111 (Other Grant/Funding Number: Ministry of Education, China); 2001BA703B02 (Other Grant/Funding Number: Ministry of Science and Technology, China); NSFC-30872173 (Other Grant/Funding Number: National Natural Science Foundation of China (NSFC)); NSFC-81102177 (Other Grant/Funding Number: National Natural Science Foundation of China (NSFC)); NSFC-81172744 (Other Grant/Funding Number: National Natural Science Foundation of China (NSFC))
Record Dates: First submitted 2007-09-21; First posted 2007-09-26 (Estimated); Last update posted 2011-12-14 (Estimated); Status verified 2011-12

CONDITIONS: Stroke
Keywords: Siblings
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum, white cells
Oversight: Data Monitoring Committee: No

SUMMARY:
The exact etiology of ischemic stroke remains unclear, because multiple genetic predispositions and environmental risk factors may be involved, and their interactions dictate the complexity. Family-based studies provide unique features in design because of their robustness to population admixture and stratification. The Fangshan / Family-based Ischemic Stroke Study In China (FISSIC) program aims to conduct a genetic pedigree study of ischemic stroke in rural communities of China.

DETAILED DESCRIPTION:
The FISSIC program is a community-based and hospital-centered genetic epidemiological study of ischemic stroke. The study design has two components: first, a family-based study of ischemic stroke pedigrees, including probands, their siblings, and their parents; second, the traditional matched case-control study of ischemic stroke cases and their unaffected spouses. Cases with confirmed ischemic stroke are included as probands; after their informed consent is obtained, their parents, siblings, and unaffected spouses are recruited and screened by using the proband-initiated contact method. Stroke status is verified at the central hospital, and the index stroke for each case is subtyped by medical records. Baseline clinical and demographic data are collected by questionnaire, and longitudinal follow-up visits are scheduled. Blood samples are collected from all enrolled participants through the three-tier prevention and health care network (village, township and county level) in the study area. The samples are sent to the central laboratory for processing, testing, and genotyping. The genotype data are then merged with the clinical, environmental, and follow-up data for analysis. Comprehensive statistical methods are applied to both family-based and case-control data to ascertain potential complex genetic and environmental factors and their interactions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of at least one ischemic stroke confirmed by the study neurologist on the basis of history, medical records, and head imaging by CT or MRI;
* At least 18 years old by the time of enrolment in the study;
* At least one full sibling or parent alive in areas nearby;
* Written informed consent by the patient or surrogate.

Exclusion Criteria:

* Diagnosis of Transient Ischemic Attack (TIA) only;
* Diagnosis of vasospasm after subarachnoid hemorrhage;
* Diagnosis of some Mendelian disorders: CADASIL, Fabry disease, MELAS, or sickle cell anaemia;
* Diagnosis of iatrogenic ischemic stroke associated with a surgical / interventional procedure such as coronary artery bypass grafting, carotid endarterectomy, or heart valve surgery;
* Diagnosis of ischemic stroke associated with autoimmune condition or endocarditis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ischemic stroke probands will be enrolled in two parts: incident cases from primary care clinic and prevalent cases from communities, and their family members will be recuited in communities.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2005-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yonghua Hu, MD, Principal Investigator — Peking University School of Public Health
Locations (1):
- The First Hospital of Fangshan District, Beijing, China

REFERENCES:
- [Background] Tang X, Hu Y, Chen D, Zhan S, Zhang Z, Dou H. The Fangshan/Family-based Ischemic Stroke Study In China (FISSIC) protocol. BMC Med Genet. 2007 Sep 10;8:60. doi: 10.1186/1471-2350-8-60. PMID 17825112